CLINICAL TRIAL: NCT06713941
Title: Study of the Management of Bone Metastases Compared to National Recommendations
Brief Title: Management of Bone Metastases
Acronym: OPTIMOS
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0905
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Bone Metastases
Keywords: Bone Metastases; bone target agent; medical care; international recommendation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bone metatases: This study involves adults with bone metastases or who have had a bone event associated with a cancer diagnosis.
  Interventions: Other: Study of the treatment

INTERVENTIONS:
Other: Study of the treatment — Intervention Description 1 * (Limit: 1000 characters) Study of prescribed treatments, treatments taken by the patients, and treatment discontinuation

SUMMARY:
Bone metastases (BM) are responsible for various bone events such as pathological fractures, spinal cord compression, preventive bone surgery, and severe bone pain requiring palliative radiotherapy management. Bone-targeted treatments, such as DENOSUMAB and bisphosphonates, are approved for preventing bone events caused by BM in patients being treated for metastatic cancer.

Clinical research on solid tumors has shown a reduction in the incidence of bone events with these treatments. Given this demonstrated effectiveness, it is important to optimize patient management by studying the characteristics of treated versus untreated patients, the incidence of bone events, and the impact of these events on patients.

A first nationwide study using EGB data (1/97th of the population) showed a low rate of management with bone-targeted treatment. Only 9% of patients with BM or a bone event associated with a cancer diagnosis received bone-targeted treatment. To validate and refine these results, we aim to replicate the protocol at Lyon Sud Hospital. Indeed, a greater amount of information will be available to answer the research question, and a number of biases can be avoided.

ELIGIBILITY:
* Inclusion Criteria * :

  -- Patients with an ICD 10 code for bone metastases: 79.5
  * And/or patients having had a skeletal event (pathological fracture; spinal cord compression; malignant hypercalcemia; bone pain and preventive orthopedic surgery or spine surgery) associated with a diagnosis of oncological pathology
  * Adult patients
  * No opposition
* Exclusion Criteria * :

  * - Patient hospitalized for a sarcoma during the pre-inclusion period and inclusion
  * Patients with a Long-Term Illiness (LTI) associated with a hospital diagnosis of Kaposi sarcoma over the same period as LTI
  * Patient with a diagnosis of pathological fracture linked to a diagnosis of osteoporosis (M80)
  * Patient under guardianship or curatorship
  * Minor patients
  * Patients not affiliated to the social security system at least 3 years before the diagnosis of MO and during the follow-up period.
  * Patient already diagnosed with known bone metastases in the previous year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves adults with bone metastases or who have had a bone event associated with a cancer diagnosis being treated at the Hospices Civils de Lyon or the University Hospital of Brest.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
. Clinical description: age at diagnosis, number of patients experiencing a bone event, number and types of comorbidities at the time of diagnosis per patient, vital status at inclusion, and date of death. | Through study completion maximum 1 year.
Age at diagnosis, age at inclusion, sex. | Through study completion maximum 1 year.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Brest University Hospital, Brest, France
  - Lyon Sud hospital, Hospices Civils de Lyon, Lyon, France